CLINICAL TRIAL: NCT02952599
Title: Non-Interventional Study on Edoxaban Treatment in Routine Clinical Practice in Patients With Venous Thromboembolism (VTE) in Korea and Taiwan
Brief Title: Edoxaban Treatment in Routine Clinical Practice in Patients With Venous Thromboembolism in Korea and Taiwan (ETNA-VTE-KOR-TWN)
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DU176b-D-A4010
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism
Keywords: Non-interventional Study; Real World Evidence; Patients with Acute VTE treated with Edoxaban; Efficacy/Safety
MeSH Terms: conditions — Venous Thromboembolism | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Edoxaban: Patients with established acute initial or recurrent VTE treated with edoxaban according to Summary of Product Characteristics (SmPC). Physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Prescribed according to approved label
  Other Names: Lixiana

SUMMARY:
According to current guidelines, duration of anticoagulant treatment after a venous thromboembolic event varies from 3 months to indefinite treatment depending on the estimated risks of venous thromboembolism (VTE) recurrence and bleeding. Current data for edoxaban are limited to a maximum treatment duration of 12 months.

Therefore, this study aims to gather further insight into efficacy (i.e. symptomatic recurrent VTE) and safety (i.e. bleeding events, liver adverse events, all-cause mortality and other drug related adverse events) of extended treatment with edoxaban up to 12 months in an unselected patient population in routine clinical practice.

DETAILED DESCRIPTION:
Edoxaban is an orally administered anticoagulant that inhibits coagulation factor Xa. It has been approved by the Ministry of Food and Drug Safety (MFDS) in Korea (date: 25th, August 2015) for the: Reduction in the risk of stroke and systemic embolism in patients with non valvular atrial fibrillation (NVAF) Treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) Reduction in the risk of recurrent DVT and PE, and by Taiwan Food and Drug Administration (TFDA) in Taiwan (date: 24th, February, 2016) for the Prevention of stroke and systemic embolism in adult patients with NVAF with one or more risk factors, such as congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, prior stroke or transient ischemic attack (TIA). Treatment of deep vein thrombosis (DVT) and pulmonary embolism (PE) following 5 to 10 days of initial therapy with a parenteral anticoagulant.

According to current guidelines, duration of anticoagulant treatment after a venous thromboembolic event varies from 3 months to indefinite treatment depending on the estimated risks of venous thromboembolism (VTE) recurrence and bleeding. Current data for edoxaban are limited to a maximum treatment duration of 12 months.

This non-interventional study aims to gather further insight into efficacy (i.e. symptomatic recurrent VTE) and safety (i.e. bleeding events, liver adverse events, all-cause mortality and other drug related adverse events) of extended treatment with edoxaban up to 12 months in approximately 350 patients in an unselected patient population in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Established acute initial or recurrent VTE
* Patients prescribed treatment with edoxaban according to package information before participation in the trial
* Written informed consent for participation in the study (ICF)
* Not simultaneously participating in any interventional study

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with established acute initial or recurrent VTE treated with edoxaban according to package information. To ensure that the physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban. Patients must have provided written informed consent for participation in the study (ICF) and should not participate simultaneously in any interventional study.
Sampling Method: Non-Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2019-10-29 (Actual); Study Completion 2019-10-29 (Actual)

PRIMARY OUTCOMES:
Rate of overall symptomatic VTE recurrence | Baseline to 12 months
  Rate of overall symptomatic VTE recurrence within 12 months
Rate of participants experiencing Real World Safety Data Events | 12 months
  Categories: VTE-related bleeding events, Drug-related adverse events, Cardiovascular Mortality, and All-cause Mortality

SECONDARY OUTCOMES:
Rate of participants taking edoxaban with symptomatic VTE recurrence | 12 months
  Rate of participants taking edoxaban with symptomatic VTE recurrence in 12 months
Rate of participants who permanently discontinued edoxaban with symptomatic VTE recurrence | 12 months
  Rate of participants who permanently discontinued edoxaban with symptomatic VTE recurrence in 12 months
Rate of participants with patient relevant outcomes | 12 months
  Patient relevant outcomes include bleeding events, strokes (ischaemic and haemorrhagic), systemic embolic events (SEE), and hospitalisations related to cardiovascular (CV) condition (including VTE related hospitalisation).

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (19):
- South Korea (9):
  - SoonChunHyang University Hospital Gumi, Gyeongsang, Gumi
  - Inje University Haeundae Paik Hospital, Busan, Haeundae-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Dong-A University Hospital, Seogu, Kwang-Jo Cho
  - Pusan National University Hospital, Busan, Seo-gu
  - Severance Hospital, Yonsei University Health System, Seoul, Seodaemun-gu
  - SoonChunHyang University Hospital Seoul, Seoul, Yongsan-gu
  - Keimyung University Dongsan Medical Center, Daegu
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju
- Taiwan (10):
  - Far Eastern Memorial Hospital, New Taipei City, Banciao District
  - Taipei Veterans General Hospital, Taipei, Beitou District
  - Chang Gung Memorial Hospital, KaoHsiung, Kaohsiung City, Niaosong District
  - Cheng Hsin General Hospital, Taipei, Pai-Tou
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Shih Lin District
  - National Taiwan University Hospital, Taipei, Zhongzheng District
  - KaoHsiung Veterans General Hospital, Kaohsiung City, Zuoying District
  - Changhua Christian Hospital, Chang-hua
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received EU and US marketing approval on or after 01 January 2014 or by the US or EU Health Authorities when regulatory submissions in both regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States and the European Union from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658